CLINICAL TRIAL: NCT01357291
Title: Evaluating New Mexico's Prison-Based Recidivism Reduction Program
Brief Title: Evaluating New Mexico's Recidivism Reduction Program
Acronym: RRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pepperdine University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPP0311F07
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Behavior
Keywords: Behavior; Drug users; Inmates
MeSH Terms: conditions — Behavior; Drug Misuse | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recidivism Reduction Program (Experimental): Inmates who were assigned to the RRP intervention.
  Interventions: Behavioral: Recidivism Reduction Program
- Business-as-usual (Active Comparator): Business-as-usual are those inmates not assigned to RRP and who receive standard inmate programming.
  Interventions: Behavioral: Business-as-usual

INTERVENTIONS:
Behavioral: Recidivism Reduction Program — Assigned to the 21-module Recidivism Reduction Program
  Other Names: RRP; Mew Mexico RRP; New MExico Recidivism Reduction Program
  Arms: Recidivism Reduction Program
Behavioral: Business-as-usual — Inmates who receive standard programming offered by New Mexico Department of Corrections prior to release.
  Other Names: Control group
  Arms: Business-as-usual

SUMMARY:
A a multi-site trial to measure the efficacy of the Recidivism Reduction Program, a prison based, twenty-one module reentry program operated by the New Mexico Department of Corrections.

DETAILED DESCRIPTION:
The New Mexico Department of Corrections Recidivism Reduction Program (RRP) is designed to provide offenders with knowledge and skills that are transferable to the community setting and to address issues that offenders will invariably face upon release to the community. Transitional coping skills, offender expectations upon release, family issues, and dealing with authority figures are a few of the challenges facing offenders upon reintegration. The Recidivism Reduction Program is aimed at preparing offenders for the potential obstacles that they may encounter upon release to the community and providing them skills to overcome the challenges that they will face. The RRP curriculum focuses on belief systems, self-esteem, and rational thinking. The RRP is a twenty-one module clinician-led program (approximately 100 hours) delivered in a group setting within months of release. Outcomes focus on measures of transition readiness, successful transition into the community, and recidivism.

ELIGIBILITY:
Inclusion Criteria:

* Inmates who have six months prior to release
* Inmates housed at one of the four experimental prisons
* Inmates willing to participate in the Recidivism Reduction Program

Exclusion Criteria:

- Housed in security Level 4 or 5

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Revocation rate | 12 months
  Percentage of subjects in each condition who are revoked from parole and returned to prison during the 12 months following their initial release.

SECONDARY OUTCOMES:
Days incarcerated | 12 months
  Total number of days incarcerated in jail or prison after initial release.
New arrests | 12 months
  Number of new arrests in the 12 months following initial release.
Self esteem | 2 months
  Inmate score on self-reported self esteem scale at two-month followup (just prior to release from prison).
Drug use self efficacy | 2 months
  Inmate score on self reported drug use self efficacy scale at 2 months followup (just prior to release from prison).
Criminal thinking | 2 months
  Inmate score on self reported criminal thinking scale at two month followup (just prior to release from prison).
Depression | 2 months
  Inmates score on self reported depression scale at 2 month followup (just prior to release from prison).
Anxiety | 2 months
  Inmates score on self reported anxiety scale at 2 month followup (just prior to release from prison).
Hostility | 2 months
  Inmates score on self reported hostility scale at 2 month followup (just prior to release from prison).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hawken, PhD, Principal Investigator — Pepperdine University
Locations (4):
- United States (4):
  - Western New Mexico Correctional Facility (WNMCF), Grants, New Mexico
  - Central New Mexico Correctional Facility (CNMCF), Los Lunas, New Mexico
  - Penitentiary of New Mexico (PNM), Santa Fe, New Mexico
  - Springer Correctional Facility (SCF), Springer, New Mexico